CLINICAL TRIAL: NCT00963209
Title: Tamoxifen Metabolism and the Impact of Tamoxifen Dose on the Level of the Active Metabolites in Endocrine Sensitive Breast Cancer Patients
Brief Title: Tamoxifen Citrate in Patients With Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr K. Zaman, Médecin associé, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000650376; CHUV-CEPO-TM; EU-20973
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: endocrine sensitive; breast cancer; tamoxifen; genotyping; phenotyping; Pharmacokinetics; Endoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tamoxifen (Experimental)
  Interventions: Drug: tamoxifen citrate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: tamoxifen citrate
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Estrogen can promote growth of endocrine sensitive breast cancer cells. Endocrine therapy with tamoxifen citrate may fight breast cancer by blocking the use of estrogen by the tumor cells. Pharmacokinetics and -genomics can have an impact on the efficacy of the treatment.

PURPOSE: This phase III trial is studying blood samples to see if the level of active metabolites of tamoxifen can be improved in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine how the increase of tamoxifen citrate dose influences the level of its major metabolites in patients with hormone-sensitive breast cancer.

Secondary

* To characterize the population pharmacokinetic profile
* To investigate the role of the other CYPs
* To assess the relation between clinical symptoms and CYP2D6 genotypes and/or active metabolites levels
* To explore the correlation between genotypes/metabolites levels and clinical outcomes in terms of tumor relapse.
* To assess the feasibility, efficacy, and safety of concentration-guided adjustment of tamoxifen citrate dosage.
* To conduct other exploratory analysis based on the eventual new data coming up in the future.

OUTLINE: Patients receive oral tamoxifen citrate (at a dose of 40 mg/day) daily for 4 months in the absence of disease progression or unacceptable toxicity.

Blood samples are collected for PK, genotyping, phenotyping, and further analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Hormone-sensitive breast cancer defined as > 10% estrogen receptor and/or > 10% progesterone receptor positivity by immunohistochemistry
* Receiving treatment with tamoxifen citrate and must be eligible for exposure to higher doses

PATIENT CHARACTERISTICS:

* No history of deep venous thrombosis or pulmonary embolism
* No history of endometrial carcinoma
* No known history of vaginal bleeding, endometriosis, endometrial hyperplasia, endometrial hypertrophy, and/or polyps
* Not pregnant or nursing
* No contraindication to tamoxifen citrate treatment
* No known allergy to midazolam or dextromethorphan

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determination of CYP2D6 genotype and determination of plasma concentrations of tamoxifen citrate and its metabolites (N-desmethyl-tamoxifen, 4-hydroxy-tamoxifen and endoxifen) under the 20 mg daily and 40 mg daily schedules | Jan 2013

SECONDARY OUTCOMES:
Patients' characteristics | prospectively
Tumor characteristics | prospectively
Cancer treatments history | prospectively
CYP3A4 (phenotype), and possibly other cytochromes involved in the metabolism and transport of drugs | prospectively
Characteristics of drug intake (date of tx initiation, current dosage and frequency, time of last intake) along with patient-reported adherence, assessed by questionnaire | prospectively
Concomitant medication | prospectively
Presence and quantitation of clinical symptoms | prospectively
Detection and classification of general comorbidities and side effects according to NCI-CTC v3.0 | prospectively
Detection of tumor relapse during the observation period of the study | prospectively

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Zaman, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Switzerland (2):
  - Hôpitaux Universitaire de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne